CLINICAL TRIAL: NCT02201706
Title: The Explore Study for the Efficacy and Safety of Multi-electrocoagulation Retinectomy in the Treatment of Retinal Re-detachment in Silicone Oil Filled Eye
Brief Title: Multi-electrocoagulation Retinectomy for Retinal Re-detachment in Silicone Oil Filled Eye
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiaofeng Lin, vice-president, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MER201407; MER201407 (Other: SunYat-senU)
Record Dates: First submitted 2014-07-15; First posted 2014-07-28 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Retinal Detachment
Keywords: Retinal detachment; silicone oil; retinectomy
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Multi-electrocoagulation retinectomy (Experimental): Retinal re-detachment in eyes with silicone oil filled,a modified surgery named Multi-electrocoagulation retinectomy will be used to re-attach the retina.
  Interventions: Procedure: Multi-electrocoagulation retinectomy

INTERVENTIONS:
Procedure: Multi-electrocoagulation retinectomy — a modified surgery named "multi-electrocoagulation retinectomy" to re-attach the retina.
  All the single surgical technique and devices involved in this modified surgery are used commonly in clinic.
  Base on this, the investigator changes the traditional sequence of these single surgical techniques, and combine them into a new surgical process.

SUMMARY:
Retinal re-detachment in silicone oil filled eye, especially in the traumatic eye, is a complex retinal detachment with poor prognosis.

In this study, the investigators try to apply a modified surgery as Multi-electrocoagulation retinectomy to reattach the retina. Here the investigators aimed to explore the safety and efficacy of this new surgical approach

DETAILED DESCRIPTION:
The relaxing retinectomy is a useful surgery for retinal re-detachment in eyes with silicone oil filled. However, it has some obvious disadvantages such as the cut of the normal retina surrounding, leaving a large area of retinal deficiency and significant exposure of retinal pigment epithelium and choroid membranes.

In this study, we try to apply a modified surgery named Multi-electrocoagulation retinectomy to re-attach the retina.

Instead of cutting through the proliferated retina directly, this new surgical approach adopts to cut the retina apart in a honeycomb shape with the help of electrocoagulation.

In this way, we not only relax the traction of the proliferative membranes, but also reserve the rest retina to cover the RPE layers.

Based on the hypothesis above, we are aiming to explore the safety and efficacy of this new surgical approach

ELIGIBILITY:
Inclusion Criteria:

1. Age 5-60 years, male or female
2. The primary retinal detachment was caused by ocular trauma, and the vitreous body is filled with silicone oil now.
3. The presence of inferior retinal re-detachment located among 3-9 o'clock.

Exclusion Criteria:

1. The primary retinal detachment was not caused by ocular trauma.
2. Location of the re-detached retina is not mainly in the inferior of the eye.
3. The fundus is unobservable because of severe corneal opacity.
4. The contralateral eye is non-functional
5. Serious heart, lung, liver and kidney dysfunction

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
retina reattachment rate | 3 months after the surgery

SECONDARY OUTCOMES:
visual acuity | Before surgery, 3days,1 week, 2 weeks, 4 weeks, 3 months and 6 months after surgery.
Intraocular pressure | Before surgery, 3days,1 week, 2 weeks, 4 weeks, 3 months and 6 months after surgery.
The degree of recurrent PVR | Before surgery, 3days,1 week, 2 weeks, 4 weeks, 3 months and 6 months after surgery.
The incidence of intraocular hemorrhage | Before surgery, 3days,1 week, 2 weeks, 4 weeks, 3 months and 6 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Lin, Dr, Principal Investigator — Zhongshan Ophthalmic Center of Sun yat-sen Universtiy
Locations (1):
- Zhongshan Ophthalmic Center of Sun yat-sen Universtiy, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Romaniuk VM. Ocular trauma and other catastrophes. Emerg Med Clin North Am. 2013 May;31(2):399-411. doi: 10.1016/j.emc.2013.02.003. PMID 23601479
- [Background] Han DP, Lewis MT, Kuhn EM, Abrams GW, Mieler WF, Williams GA, Aaberg TM. Relaxing retinotomies and retinectomies. Surgical results and predictors of visual outcome. Arch Ophthalmol. 1990 May;108(5):694-7. doi: 10.1001/archopht.1990.01070070080039. PMID 2334327
- [Background] de Silva DJ, Kwan A, Bunce C, Bainbridge J. Predicting visual outcome following retinectomy for retinal detachment. Br J Ophthalmol. 2008 Jul;92(7):954-8. doi: 10.1136/bjo.2007.131540. Epub 2008 Jun 12. PMID 18556423
- [Derived] Jiang Z, Qiu S, Lou B, Lin M, Tan J, Lin X. Radial Retinotomies with Endodiathermy for Severe Proliferative Vitreoretinopathy: Short-Term Results. J Ophthalmol. 2016;2016:2594574. doi: 10.1155/2016/2594574. Epub 2016 Feb 28. PMID 27022477